CLINICAL TRIAL: NCT00195182
Title: Psychosocial Determinants of Medication Adherence in Hypertensive African Americans
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Other Study IDs: 0302006001
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2008-05-21 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension
Keywords: Hypertension; African-American; Perceived Racism; Psychological Stress; Medication Adherence
MeSH Terms: conditions — Hypertension; Stress, Psychological; Medication Adherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1. No intervention: This group received follow-up every 2-months for one year. Follow-up included questions about their blood pressure and how well they had been able to adhere to their medication goal.
  Interventions: Behavioral: Self affirmation and positive affect induction vs. control
- 2. Experimental: This group received follow-up every 2-months for one year. Follow-up included questions about their blood pressure and how well they had been able to engage adhere to their medication goal. The intervention included receiving an additional educational workbook about using positive affect and self affirmation, as well as participating in using positive affect and self-affirmation to motivate behavior change, which in this case was to increase their physical activity level.
  Interventions: Behavioral: Self affirmation and positive affect induction vs. control

INTERVENTIONS:
Behavioral: Self affirmation and positive affect induction vs. control — During the physical activity goal setting process, subjects were randomly assigned to either the control or the intervention group. The intervention included receiving an additional educational workbook about using positive affect and self affirmation, as well as participating in using positive affect and self-affirmation to motivate behavior change, which in this case was to increase their medication adherence. Patient also received small token gifts to remind them of their participation in the study and to induce positive affect. The control group also set a physical activity goal and received the same follow-up, but did not participate in the positive affect and self-affirmation portion.

SUMMARY:
The specific aims for this study are:

1. To examine the relationship between perceived racism and medication adherence among hypertensive African-American patients.
2. To determine if psychological stress and depression mediate the relationship between perceived racism and medication adherence.

DETAILED DESCRIPTION:
Achieving and maintaining recommended blood pressure goals in hypertensive African Americans is paramount to addressing racial disparities in hypertension-related morbidity and mortality. Because antihypertensive therapy is the cornerstone of hypertension management, good medication adherence is the key to adequate blood pressure control. Successful approaches to racial disparities must address how to increase adherence to anti-hypertensive medications.

Adherence to anti-hypertensive medications is likely multifactorial, and not solely related to SES or access to medical care. Psychosocial factors such as stress and depression have been implicated as important determinants of medication adherence. However, little is known about how other psychosocial factors such as perceived racism impact anti-hypertensive medication adherence. Understanding these relationships may assist in the development of targeted strategies to achieve good medication adherence in hypertensive patients.

The objective is to understand the relationships between perceived racism and medication adherence, while examining the role of depression, psychological stress, and self-efficacy in a population of hypertensive African-American patients. 262 African American adult hypertensive patients will be recruited from an urban academic general medicine practice. Baseline data collection will include assessments of demographics and socioeconomic status, clinical history and hypertension characteristics, depressive symptoms, perceived stress, and medication adherence. Patients will be followed for 1 year, when final evaluations will take place, including assessment of hypertension, stress, depression, medication adherence and level of perceived racism (measured by a validated instrument). The primary outcome is the change in medication adherence scores from baseline to 12 months. Statistical models will be developed to determine if level of perceived racism is associated with medication adherence, and whether stress and depression play a role in this relationship.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be self-identified as African American.
2. All patients must be aged 18 years or older.
3. All patients must be diagnosed as having hypertension (for this project, hypertension will be defined according to the widely accepted criteria of the 6th Joint National Committee Guidelines on Prevention, Detection, Evaluation and Treatment of Hypertension, specifically a systolic blood pressure >140 mm hg or a diastolic blood pressure >90 mm hg) or if patients are taking any prescribed anti-hypertensive medication.
4. Patients must be able to provide informed consent in English.

Exclusion Criteria:

1. Patients who are unable to walk several blocks for any reason.
2. Patients who refused to participate.
3. Patients who are unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive African Americans
Sampling Method: Non-Probability Sample
Enrollment: 262 (Estimated)
Dates: Start 2003-09; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
To evaluate intervention of induced positive affect and induced self-affirmation will increase medication adherence among African-American hypertensive patients. | every two months for one year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph E Ravenell, MD, MS, Principal Investigator — University of Texas Southwestern Medical Center; Mary E Charlson, MD, Study Director — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital-Weill Medical College, New York, New York, United States

REFERENCES:
- [Background] Ravenell JE, Charlson ME. Stressed out: Definitions of stress among hypertensive African American men. Journal of General Internal Medicine 20(S1):128, 2005.